CLINICAL TRIAL: NCT02675933
Title: What Factors Effect Parental Satisfaction During Their Visit to a Pediatric Emergency Department Among Parents of Children With Autism?
Brief Title: Satisfaction Rates Among Parents of Children With Autism in the ED
Acronym: ASD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Seton IRB administratively closed this study on January 6, 2017
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-15-162
Record Dates: First submitted 2016-01-31; First posted 2016-02-05 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): The control arm participants will receive only a satisfaction survey once disposition is determined by the physician provider. The satisfaction survey will be collected by the research associated and kept in a protected location, along with all other study materials.
  All patients will receive standard of care, which at this institution is the help of Child Life Specialists, when they are available and requested by the physician. Physicians will be instructed to request Child Life Specialists with the same discretion as with all patients.
- Questionnaire (Active Comparator): Participants who are randomized to the questionnaire arm will receive a patient-centered questionnaire at the beginning of their visit. This single page document will ask questions about their child including, but not limited to, diagnoses, suggestions for distraction, sensory issues that may affect their visit, and method to best administer medications. The research associate will ask them to fill it out to the best of their ability and will collect the questionnaire prior to a physician provider seeing the patient. At least one physician provider must review the questionnaire prior to seeing the patient.
  Once disposition is determined, the satisfaction survey will be distributed by the research associate along with an envelope for the parent to seal their survey within.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — There will be a single page document, a patient-centered questionnaire, distributed to parents of study participants who have been randomized to the intervention arm.
  Arms: Questionnaire

SUMMARY:
This study is a randomized controlled trial utilizing a patient-centered questionnaire distributed to parents of children with autism. The study arm will receive the questionnaire and will be compared to the control arm, which will receive standard of care. The results of satisfaction surveys will be the primary endpoint of this study.

DETAILED DESCRIPTION:
This study is a randomized controlled trial utilizing a patient-centered questionnaire distributed to parents of children with autism. Potential study participants will be identified during the triage process through medical history taking, which is routine for the triage process at this institution. The triage nurse will be educated to alert a research associate if a patient with one of our qualifying diagnoses is identified. This study will include patients aged 2-18 with parental report of a diagnosis of (1) Autism, (2) Autism Spectrum Disorder, (3) Pervasive Developmental Disorder, (4) Childhood Disintegrative Disorder, or (5) Sensory Integration Disorder. All patients whose caregiver is fluent and literate in either English or Spanish will be included.

Research associates will then attempt to obtain consent from the parent. If consent is obtained, the research associate will then attempt to obtain assent from patients aged > 6 years. If the research associate feels the child is unable to assent based on their developmental capabilities, the research associate will then indicate this on the assent form and sign in the space provided for the research associate.

Once consent and assent, if applicable, are obtained, the research associate will then select an envelope from the top of a pre-randomized stack. The contents of the envelope will either contain a questionnaire and satisfaction survey for the intervention arm, or simply a satisfaction survey if in the control arm.

If the intervention arm is selected, the research associate will then distribute the questionnaire to the parent and ask them to fill it out to the best of their ability. The research associate will then return to collect the questionnaire and one of the physician providers caring for the patient must review the questionnaire prior to seeing the patient. This hospital is a teaching institution and physician providers may include residents, fellows, and attendings.

Once reviewed, the physician provider will sign at the bottom of the questionnaire and proceed with the encounter. Multiple providers, including nursing staff and clinical assistants may review the questionnaire as well, which will be kept on the paper chart.

When the patient's disposition is determined, the research associate will distribute the satisfaction survey and an envelope for the survey to be sealed within once completed by the parent. The satisfaction survey, along with the questionnaire and any other study documents, will be collected and placed in the envelope. The envelopes will be stored in a badge-access protected office inside of a locked cabinet behind a password protected door. Only fellows, attendings, and a few fellowship-associated and research-associated providers have access to this office.

ELIGIBILITY:
Inclusion Criteria:

* aged 2 to 18 years
* parent/caregiver is fluent and literate in either English or Spanish
* parental report of a diagnosis of (1) autism, (2) autism spectrum disorder, (3) pervasive developmental disorder, (4) childhood disintegrative disorder, (5) sensory integration disorder

Exclusion Criteria:

* triage level 1
* physician provider unable to review questionnaire prior to seeing the patient

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Yee, MD, Principal Investigator — Pediatric Emergency Medicine Fellow
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Jo H, Schieve LA, Rice CE, Yeargin-Allsopp M, Tian LH, Blumberg SJ, Kogan MD, Boyle CA. Age at Autism Spectrum Disorder (ASD) Diagnosis by Race, Ethnicity, and Primary Household Language Among Children with Special Health Care Needs, United States, 2009-2010. Matern Child Health J. 2015 Aug;19(8):1687-97. doi: 10.1007/s10995-015-1683-4. PMID 25701197
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193

RESULTS

PARTICIPANT FLOW:
Groups:
- Questionnaire: Participants who are randomized to the questionnaire arm will receive a patient-centered questionnaire at the beginning of their visit. This single page document will ask questions about their child including, but not limited to, diagnoses, suggestions for distraction, sensory issues that may affect their visit, and method to best administer medications. The research associate will ask them to fill it out to the best of their ability and will collect the questionnaire prior to a physician provider seeing the patient. At least one physician provider must review the questionnaire prior to seeing the patient.
  Once disposition is determined, the satisfaction survey will be distributed by the research associate along with an envelope for the parent to seal their survey within.
  Questionnaire: There will be a single page document, a patient-centered questionnaire, distributed to parents of study participants who have been randomized to the intervention arm.
Period: Overall Study
Arm/Group | Standard of Care | Questionnaire
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Questionnaire | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 31 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.32 [2 to 15] | 8.72 [2 to 17] | 8.52 [2 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction Scores
Description: Parental satisfaction as rated on a Likert Scale (1-5) with higher number/scores (5) meaning a better outcome.
Time Frame: through study completion, 1 day (clinic visit)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard of Care | Questionnaire
Number analyzed (Participants) | 32 | 31
score on a scale | 4.1 [1 to 5] | 4.5 [1 to 5]

ADVERSE EVENTS:
Time Frame: through study completion, 1 day (clinic visit)
Description: This study involved collection of patient and parent preference data through the use of a questionnaire. There were no medications or devices involved in the study.
Arm/Group | Standard of Care | Questionnaire
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=32) | Questionnaire (N=31)
Data breach (Investigations) | 0 (0) | 0 (0) — Data breach is only risk with a questionnaire

LIMITATIONS AND CAVEATS:
No final reported analysis. Study terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No